CLINICAL TRIAL: NCT02927405
Title: Combination of Preoperative Gabapentin and TAP Blocks in Decreasing Postoperative Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not get the study to take off, did not recruit any subjects, and then closed the study.
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Shantha Ganesan, Director, Pain Medicine, State University of New York - Downstate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 926072
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain
Keywords: gabapentin; TAP block
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAP Block plus placebo (Placebo Comparator): Patients will only receive a TAP block procedure and then morphine consumption will be recorded.
  Interventions: Procedure: TAP Block
- TAP Block plus gabapentin (Experimental): Patients will receive a TAP block procedure and take pre-operative oral Gabapentin and morphine consumption will me recorded after surgery.
  Interventions: Drug: Gabapentin; Procedure: TAP Block

INTERVENTIONS:
Drug: Gabapentin — anticonvulsant drug that is used for neuropathic pain.
  Other Names: Neurontin
  Arms: TAP Block plus gabapentin
Procedure: TAP Block — a procedure done anesthetize the anterior abdominal wall

SUMMARY:
There is an increasing trend on decreasing narcotic use and maximizing efficiency in the perioperative care. There are no studies that have compared a TAP block versus a TAP block plus gabapentin for laparoscopic procures.This study will investigate if taking gabapentin and receiving a TAP block decrease post-operative morphine consumption. It will be a randomized controlled, double blind study, with 130 patients between 18-60 years; that will undergo laparoscopic GYN procedures. Secondary outcomes will look at the incidence of nausea, vomiting, and VAS (verbal analog scale) scores. This combination may be helpful because gabapentin will be used to decrease visceral and central pain, and TAP block will decrease somatic pain. Performing a multimodal approach may decrease narcotic consumption, adverse effects and improve pain management.

ELIGIBILITY:
Inclusion Criteria:

* female
* receiving laparoscopic GYN procedure
* between 18-60

Exclusion Criteria:

* are already taking gabapentin
* have diabetic neuropathy
* have a chronic pain syndrome
* take opioids at home
* are pregnant
* have kidney disease
* have an allergy to morphine

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-04 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative morphine consumption | 24 hours after surgery.
  Total amount of morphine the patient need to control post-operative pain

SECONDARY OUTCOMES:
VAS Scores | 24 hours after surgery
  Visual analog scale that rates a patient's pain

OTHER OUTCOMES:
Incidence of nausea and vomiting | 24 hours after surgery
  How many times the patient reported nausea, and how many times they vomitted.

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Downstate Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No